CLINICAL TRIAL: NCT00815022
Title: Influence of Anesthetic Temperature on Cephalad Sensory Blockade With Spinal Anesthesia for Cesarean Delivery
Brief Title: Influence of Anesthetic Temperature on Cephalad Sensory Blockade With Spinal Anesthesia
Acronym: ATOCEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Fu Zhou Wang, Dr, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMU-200812-MZ32; NJFY0812009
Record Dates: First submitted 2008-12-26; First posted 2008-12-29 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Cesarean Delivery
Keywords: Temperature; Spinal anesthesia; Cesarean section; Cephalad sensory blockade; Regional anesthesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Active Comparator): Mixture of anesthetic including hyperbaric bupivacaine 12 mg, fentanyl 10 microg and morphine 200 microg, with the temperature of 20 degree celsius
  Interventions: Drug: bupivacaine/fentanyl/morphine
- 2 (Experimental): Mixture of anesthetic including hyperbaric bupivacaine 12 mg, fentanyl 10 microg and morphine 200 microg, with the temperature of 10 degree celsius
  Interventions: Drug: bupivacaine/fentanyl/morphine
- 3 (Experimental): Mixture of anesthetic including hyperbaric bupivacaine 12 mg, fentanyl 10 microg and morphine 200 microg, with the temperature of 15 degree celsius
  Interventions: Drug: bupivacaine/fentanyl/morphine
- 4 (Experimental): Mixture of anesthetic including hyperbaric bupivacaine 12 mg, fentanyl 10 microg and morphine 200 microg, with the temperature of 25 degree celsius
  Interventions: Drug: bupivacaine/fentanyl/morphine
- 5 (Experimental): Mixture of anesthetic including hyperbaric bupivacaine 12 mg, fentanyl 10 microg and morphine 200 microg, with the temperature of 30 degree celsius
  Interventions: Drug: bupivacaine/fentanyl/morphine
- 6 (Experimental): Mixture of anesthetic including hyperbaric bupivacaine 12 mg, fentanyl 10 microg and morphine 200 microg, with the temperature of 35 degree celsius
  Interventions: Drug: bupivacaine/fentanyl/morphine

INTERVENTIONS:
Drug: bupivacaine/fentanyl/morphine — Hyperbaric bupivacaine 12 mg, fentanyl 10 microg and morphine 200 microg

SUMMARY:
Several factors influence the extension of anesthetic mixture during spinal anesthesia including anesthetic gravity, body position, drug volume, and drug-delivering velocity. However, the effect of temperature of anesthetic mixture on the cephalad sensory blockade is hitherto unknown. The investigators hypothesized that different temperatures of the anesthetic mixture had different velocity of extension after spinal anesthesia. In addition, previous studies suggest that parturients have relative higher sensitivity to temperature. Herein the investigators proposed that the temperature of anesthetic mixture had more extensive effect on the cephalad sensory blockade with spinal anesthesia for cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous women
2. > 18 years and < 45 years

Exclusion Criteria:

1. Allergy to opioids, a history of the use of centrally-acting drugs of any sort, chronic pain and psychiatric diseases records
2. Participants younger than 18 years or older than 45 years
3. Those who were not willing to or could not finish the whole study at any time
4. Alcohol addictive or narcotic dependent patients
5. Subjects with a nonvertex presentation
6. Diagnosed diabetes mellitus and pregnancy-induced hypertension
7. Twin gestation and breech presentation
8. Pregnant fever

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2008-12; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum cephalad sensory blockade to pinprick, cold and touch | From the delivery of anesthetic mixture to 15 min immediate after spinal anesthesia

SECONDARY OUTCOMES:
Velocity of the sensory blockade at identical body position | From the delivery of anesthetic mixture to 15 min immediate after spinal anesthesia
The total dose of phenylephrine required to maintain baseline arterial blood pressure | From the delivery of anesthetic mixture to 25 min after spinal anesthesia
Time interval of the occurrence of the hypotension | From the delivery of the anesthetic mixture to 25 min after spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China